CLINICAL TRIAL: NCT04075318
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of UBITh® PD Immunotherapeutic Vaccine (UB-312) in Healthy Participants and Participants With Parkinson's Disease
Brief Title: Study of UB-312 in Healthy Participants and Parkinson's Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Neuroscience Ltd. (Industry)
Collaborators: Centre for Human Drug Research, Netherlands (Other); Worldwide Clinical Trials (Other); Vaxxinity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UB-312-101
Record Dates: First submitted 2019-08-05; First posted 2019-08-30 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Disease; Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part A: UB-312 40 mcg (Experimental): UB-312 40 mcg by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: UB-312
- Part A: UB-312 100 mcg (Experimental): UB-312 100 mcg by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: UB-312
- Part A: UB-312 40/300 mcg (Experimental): UB-312 40 mcg at Week 1 and 300 mcg at Weeks 5 and 13 by intramuscular injection
  Interventions: Biological: UB-312
- Part A: UB-312 300 mcg (Experimental): UB-312 300 mcg by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: UB-312
- Part A: UB-312 40/1000 mcg (Experimental): UB-312 40 mcg at Week 1 and 1000 mcg at Weeks 5 and 13 by intramuscular injection
  Interventions: Biological: UB-312
- Part A: UB-312 1000 mcg (Experimental): UB-312 1000 mcg by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: UB-312
- Part A: UB-312 2000 mcg (Experimental): UB-312 2000 mcg by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: UB-312
- Part A: Placebo (Placebo Comparator): Placebo by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: Placebo
- Part B: UB-312 300/100 mcg (Experimental): UB-312 300 mcg at Week 1 and 100 mcg at Weeks 5 and 13 by intramuscular injection
  Interventions: Biological: UB-312
- Part B: UB-312 300 mcg (Experimental): UB-312 300 mcg at Weeks 1, 5 and 13 by intramuscular injection
  Interventions: Biological: UB-312
- Part B: Placebo (Placebo Comparator): Placebo by intramuscular injection at Weeks 1, 5 and 13
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UB-312 — A synthetic peptide-based vaccine
  Arms: Part A: UB-312 100 mcg; Part A: UB-312 1000 mcg; Part A: UB-312 2000 mcg; Part A: UB-312 300 mcg; Part A: UB-312 40 mcg; Part A: UB-312 40/1000 mcg; Part A: UB-312 40/300 mcg; Part B: UB-312 300 mcg; Part B: UB-312 300/100 mcg
Biological: Placebo — Matching placebo
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
This is a 44-week, randomized, placebo-controlled, double-blind, single-center, phase 1 clinical trial consisting of a dose-escalation Part A study in healthy participants, followed by a Part B in participants with Parkinson's disease with a selected doses from Part A.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1 study to determine the safety, tolerability, and immunogenicity of UB-312 in healthy participants and in participants with Parkinson's disease (PD). UB-312 is a UBITh®-enhanced synthetic peptide-based vaccine and may provide an active immunotherapy option for treating synucleinopathies including the most prevalent form, PD.

The study consists of two parts. Part A of the study with healthy participants will consist of dose escalation and cohort staggering for up to seven planned dose levels or placebo. Part B of the study will consist of two cohorts of participants with Parkinson's disease (PD). Dosing for Part B will be based on safety, tolerability and immunogenicity from Part A. All eligible participants will be enrolled in a 44-week study consisting of 20 weeks of treatment and 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40 to 85 years old, inclusive at screening
* Expected to be able to undergo all study procedures
* Other inclusion criteria apply

For Part B only:

* A diagnosis of PD, confirmed by a neurologist
* Hoehn &Yahr Stage ≤ III at Screening
* Stable treatment of permitted antiparkinsonian medications from 30 days prior to first study drug administration or 60 days for MAO-B inhibitors, and expected to remain stable throughout the study

Exclusion Criteria:

* Clinically significant abnormalities, as judged by the investigator
* History of medical, neurological or psychiatric conditions which in the opinion of the investigator may compromise participant's safety or scientific value of the study
* Acute or chronic infection as judged by the investigator, for positive human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV)
* History or evidence of an autoimmune disorder
* History of anergy.
* Participated/participating in any clinical trial with monoclonal antibodies or vaccines directed at aSyn
* Other exclusion criteria apply

For Part B only:

* Other known or suspected cause of Parkinsonism other than idiopathic PD
* History or evidence at Screening of PD-related freezing episodes, falls, or orthostatic hypotension
* Dopamine transporter single-photon emission computerized tomography scan (DaTscan) inconsistent with dopamine transporter deficit.
* Clinically significant neurological disease other than PD

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Vaxxinity, Inc.
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CY, Walfield AM. Site-specific peptide vaccines for immunotherapy and immunization against chronic diseases, cancer, infectious diseases, and for veterinary applications. Vaccine. 2005 Mar 18;23(17-18):2049-56. doi: 10.1016/j.vaccine.2005.01.007. PMID 15755569
- [Background] Wang CY, Finstad CL, Walfield AM, Sia C, Sokoll KK, Chang TY, Fang XD, Hung CH, Hutter-Paier B, Windisch M. Site-specific UBITh amyloid-beta vaccine for immunotherapy of Alzheimer's disease. Vaccine. 2007 Apr 20;25(16):3041-52. doi: 10.1016/j.vaccine.2007.01.031. Epub 2007 Jan 19. PMID 17287052
- [Background] Wang CY, Wang PN, Chiu MJ, Finstad CL, Lin F, Lynn S, Tai YH, De Fang X, Zhao K, Hung CH, Tseng Y, Peng WJ, Wang J, Yu CC, Kuo BS, Frohna PA. UB-311, a novel UBITh(R) amyloid beta peptide vaccine for mild Alzheimer's disease. Alzheimers Dement (N Y). 2017 Apr 14;3(2):262-272. doi: 10.1016/j.trci.2017.03.005. eCollection 2017 Jun. PMID 29067332
- [Result] Eijsvogel P, Misra P, Concha-Marambio L, Boyd JD, Ding S, Fedor L, Hsieh YT, Sun YS, Vroom MM, Farris CM, Ma Y, de Kam ML, Radanovic I, Vissers MFJM, Mirski D, Shareghi G, Shahnawaz M, Singer W, Kremer P, Groeneveld GJ, Yu HJ, Dodart JC. Target engagement and immunogenicity of an active immunotherapeutic targeting pathological alpha-synuclein: a phase 1 placebo-controlled trial. Nat Med. 2024 Sep;30(9):2631-2640. doi: 10.1038/s41591-024-03101-8. Epub 2024 Jun 20. PMID 38902546
- [Result] Yu HJ, Thijssen E, van Brummelen E, van der Plas JL, Radanovic I, Moerland M, Hsieh E, Groeneveld GJ, Dodart JC. A Randomized First-in-Human Study With UB-312, a UBITh(R) alpha-Synuclein Peptide Vaccine. Mov Disord. 2022 Jul;37(7):1416-1424. doi: 10.1002/mds.29016. Epub 2022 Apr 15. PMID 35426173

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A: UB-312 40 mcg | Part A: UB-312 100 mcg | Part A: UB-312 40/300 mcg | Part A: UB-312 300 mcg | Part A: UB-312 40/1000 mcg | Part A: UB-312 1000 mcg | Part A: UB-312 2000 mcg | Part A: Placebo | Part B: UB-312 300/100 mcg | Part B: UB-312 300 mcg | Part B: Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 7 | 6
Completed | 6 | 6 | 5 | 6 | 0 | 0 | 0 | 5 | 6 | 7 | 6
Not Completed | 0 | 0 | 1 | 0 | 6 | 6 | 6 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: UB-312 40 mcg | Part A: UB-312 100 mcg | Part A: UB-312 40/300 mcg | Part A: UB-312 300 mcg | Part A: UB-312 40/1000 mcg | Part A: UB-312 1000 mcg | Part A: UB-312 2000 mcg | Part A: Placebo | Part B: UB-312 300/100 mcg | Part B: UB-312 300 mcg | Part B: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 7 | 6 | 70
Age, Continuous [Mean (Full Range); unit: years] | 72.5 [62 to 79] | 65.0 [49 to 79] | 68.5 [49 to 77] | 60.0 [46 to 77] | 65.0 [44 to 85] | 68.3 [64 to 73] | 72.0 [64 to 80] | 64.6 [41 to 76] | 67.4 [44 to 83] | 63.4 [50 to 75] | 61.0 [51 to 73] | 66.1 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 4 | 2 | 1 | 4 | 4 | 1 | 2 | 1 | 29
  Male | 4 | 2 | 2 | 2 | 4 | 5 | 2 | 4 | 6 | 5 | 5 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Other: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other: Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Other: White | 6 | 5 | 6 | 6 | 5 | 6 | 5 | 7 | 7 | 7 | 6 | 66
  Other: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other: Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 7 | 6 | 70

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: Number of AEs will be assessed
Time Frame: 44 weeks
Measure: Number; unit: TEAEs
Arm/Group | Part A: UB-312 40 mcg | Part A: UB-312 100 mcg | Part A: UB-312 40/300 mcg | Part A: UB-312 300 mcg | Part A: UB-312 40/1000 mcg | Part A: UB-312 1000 mcg | Part A: UB-312 2000 mcg | Part A: Placebo | Part B: UB-312 300/100 mcg | Part B: UB-312 300 mcg | Part B: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 7 | 6
TEAEs | 22 | 31 | 25 | 31 | 24 | 17 | 18 | 25 | 59 | 42 | 20

2. Primary Outcome: Immunogenicity of UB-312 as Determined by Anti-aSyn Antibodies in Blood
Description: Number of Participants with Anti-aSyn Antibodies in Blood from Weeks 1 through 45.
Time Frame: 44 weeks
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: UB-312 40 mcg | Part A: UB-312 100 mcg | Part A: UB-312 40/300 mcg | Part A: UB-312 300 mcg | Part A: UB-312 40/1000 mcg | Part A: UB-312 1000 mcg | Part A: UB-312 2000 mcg | Part A: Placebo | Part B: UB-312 300/100 mcg | Part B: UB-312 300 mcg | Part B: Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 0 | 0 | 0 | 5 | 6 | 7 | 6
Participants | 5 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 5 | 7 | 0

3. Primary Outcome: Immunogenicity of UB-312 as Determined by Anti-aSyn Antibodies in CSF
Description: Number of Participants with Anti-aSyn Antibodies in CSF from Weeks 1 through 45.
Time Frame: 44 weeks
Population: per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: UB-312 40 mcg | Part A: UB-312 100 mcg | Part A: UB-312 40/300 mcg | Part A: UB-312 300 mcg | Part A: UB-312 40/1000 mcg | Part A: UB-312 1000 mcg | Part A: UB-312 2000 mcg | Part A: Placebo | Part B: UB-312 300/100 mcg | Part B: UB-312 300 mcg | Part B: Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 0 | 0 | 0 | 5 | 6 | 7 | 6
Participants | 1 | 4 | 3 | 6 | 0 | 0 | 0 | 0 | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the length of the participants enrollment in the study which was 44 weeks.
Description: Definition does not differ.
Arm/Group | Part A: UB-312 40 mcg | Part A: UB-312 100 mcg | Part A: UB-312 40/300 mcg | Part A: UB-312 300 mcg | Part A: UB-312 40/1000 mcg | Part A: UB-312 1000 mcg | Part A: UB-312 2000 mcg | Part A: Placebo | Part B: UB-312 300/100 mcg | Part B: UB-312 300 mcg | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/7 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 3/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 6/6 | 6/6 | 6/6 | 5/6 | 8/8 | 7/7 | 7/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: UB-312 40 mcg (N=6) | Part A: UB-312 100 mcg (N=6) | Part A: UB-312 40/300 mcg (N=6) | Part A: UB-312 300 mcg (N=6) | Part A: UB-312 40/1000 mcg (N=6) | Part A: UB-312 1000 mcg (N=6) | Part A: UB-312 2000 mcg (N=6) | Part A: Placebo (N=8) | Part B: UB-312 300/100 mcg (N=7) | Part B: UB-312 300 mcg (N=7) | Part B: Placebo (N=6)
Hospital Acquired Pneumonia (HAP) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unprovoked Deep Venous Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: UB-312 40 mcg (N=6) | Part A: UB-312 100 mcg (N=6) | Part A: UB-312 40/300 mcg (N=6) | Part A: UB-312 300 mcg (N=6) | Part A: UB-312 40/1000 mcg (N=6) | Part A: UB-312 1000 mcg (N=6) | Part A: UB-312 2000 mcg (N=6) | Part A: Placebo (N=8) | Part B: UB-312 300/100 mcg (N=7) | Part B: UB-312 300 mcg (N=7) | Part B: Placebo (N=6)
Eye Disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
General Disorders and Administration Site Conditions (General disorders) | 5 (9) | 4 (9) | 4 (7) | 6 (13) | 4 (6) | 6 (11) | 5 (7) | 5 (6) | 4 (8) | 2 (4) | 3 (5)
Immune System Disorders (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and Infestations (Immune system disorders) | 1 (1) | 4 (5) | 3 (5) | 2 (3) | 3 (3) | 2 (2) | 3 (3) | 5 (8) | 4 (9) | 5 (10) | 1 (1)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 2 (3)
Muscoloskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4) | 1 (1) | 4 (5) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (8) | 2 (2) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 4 (8) | 3 (7) | 3 (6) | 3 (6) | 3 (9) | 2 (2) | 4 (4) | 5 (7) | 6 (14) | 7 (13) | 4 (4)
Psychiatric Disorders (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Renal and Urinary Disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Surgical and Medical Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular Disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT04075318/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT04075318/SAP_001.pdf